CLINICAL TRIAL: NCT02411526
Title: An Open-Label, Multiple Dose, Safety and Pharmacokinetic Trial With Injectable ZX003 (Risperidone-SABER®) Compared to Risperdal® Consta® in Patients With Chronic, Stable Schizophrenia or Schizoaffective Disorder
Brief Title: Safety and PK Trial With Injectable ZX003 (Risperidone-SABER®) Compared to Risperdal® Consta® in Stable Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZX003-1401
Record Dates: First submitted 2015-03-16; First posted 2015-04-08 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2015-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 60 mg of ZX003 administered 4 times (every 4 weeks)
  Interventions: Drug: ZX003 (Risperidone-SABER®)
- Cohort 2 (Experimental): 90 mg of ZX003 administered 4 times (every 4 weeks)
  Interventions: Drug: ZX003 (Risperidone-SABER®)
- Cohort 3 (Experimental): 120 mg of ZX003 administered 4 times (every 4 weeks)
  Interventions: Drug: ZX003 (Risperidone-SABER®)
- Cohort 4 (Active Comparator): Risperdal Consta administered 5 times (once every 2 weeks) NOTE: Oral risperidone 2 mg will be given with the first injection of Risperdal Consta and continued for 3 weeks (and then discontinued) to ensure adequate therapeutic plasma concentrations from Risperdal Consta.
  Interventions: Drug: Risperdal Consta; Drug: Oral Risperidone

INTERVENTIONS:
Drug: ZX003 (Risperidone-SABER®) — ZX003 administered as a SC injection
  Other Names: Relday
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Risperdal Consta — Risperdal Consta administered as a IM injection
  Other Names: risperidone
  Arms: Cohort 4
Drug: Oral Risperidone — Oral Risperidone given to ensure adequate therapeutic plasma concentrations from Risperdal Consta
  Other Names: risperdal
  Arms: Cohort 4

SUMMARY:
This is an open-label, multiple dose, PK and safety study in patients with chronic, stable schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Approximately 75 male and female patients with schizophrenia or schizoaffective disorder on antipsychotic maintenance medication will be enrolled into the study. There will be 4 planned cohorts of 14 patients per cohort.

In Cohorts 1-3, patients' planned participation in the study is for a total of approximately 22 weeks, including a Screening period of up to 35 days, and a study treatment period of 120 days (including follow-up).

In Cohort 4 planned participation in the study is for a total of approximately 18 weeks including a Screening period of up to 35 days and a study treatment of 92 days (including follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 - 60 years of age, inclusive.
2. Diagnosis of schizophrenia, or schizoaffective disorder as per DSM-V criteria in the past 6 months or more, dependent on diagnosis.
3. Currently on maintenance antipsychotic medication (ie, patients treated with antipsychotic medication with stable doses in the 4 weeks prior to Screening and no psychosis-related dose changes in the 8 weeks prior to Screening).
4. Body Mass Index (BMI) ≥20 and ≤40 kg/m2.
5. Female patients who are non-childbearing potential (surgically sterile [hysterectomy]) or post-menopausal ≥2 years; or non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (hormonal contraception, abstinence, diaphragm with spermicide, condom with spermicide, or intrauterine device) from Screening until the End-of-Study visit.
6. No clinically significant abnormal laboratory values.
7. No clinically significant findings in the 12-lead ECG.
8. No clinically significant findings from a vital signs measurement.
9. Be informed of the nature of the study and give written consent prior to initiating any study procedure.

Exclusion Criteria:

1. Unwilling to provide genotyping (phenotyping) sample for CYP2D6.
2. Have known or suspected carcinoma.
3. Have known presence or history of renal or hepatic insufficiency.
4. Have known history, hypersensitivity or clinically significant idiosyncratic reaction to risperidone, paliperidone, and/or any other drug substance with similar activity.
5. Have a history of alcohol or drug-dependence as per DSM-V criteria during the 6-month period immediately prior to Screening.
6. Have a history of epilepsy or risk of having seizures.
7. Are pregnant, lactating, or likely to become pregnant during the study.
8. Have taken an antipsychotic depot product (including investigational products) within the 60 days prior to Screening.
9. Participated in another clinical trial or received an investigational product within 30 days prior to Screening.
10. Have a positive alcohol breathalyzer test at Screening or Admission.
11. Have a positive Screening test for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
12. Have a positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines (unless prescribed), cannabinoids, etc.) at Screening or Admission.
13. Excessive use of caffeine-containing beverages exceeding 500 mg caffeine/day (5 cups of coffee).
14. Use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to Admission.
15. Excessive smoking, defined as smoking more than 2 packs of cigarettes (or 5 cigars) per day for 1 year or greater.
16. Donation of blood (>500 mL) or blood products within 2 months (56 days) prior to Admission.
17. Have used any concomitant medications significantly impacting CYP2D6 (moderate and strong inducers/inhibitors),within 14 days or 5 half-lives (whichever is longer) prior to Admission. Medications judged to not interact with risperidone may be continued at the discretion of the Investigator and in accordance with the protocol requirements for tapering and washout.
18. Are unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study.
19. Are unlikely to comply with the protocol requirements, instructions and study- related restrictions (eg, uncooperative attitude, inability to return for out-patient visits or improbability of completing the clinical study).
20. Are unable to tolerate the Oral Risperidone Challenge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
PK profile of ZX003 determined by C max, T max, C min, AUC (0-24h), AUC (0-tau), C avg | Day 1 through day 120

SECONDARY OUTCOMES:
Safety and tolerability of ZX003 as measured by assessing adverse events. | Day 1 through day 120
Safety and tolerability of ZX003 as measured by assessing laboratory values. | Day 1 through day 120

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, PhD, Principal Investigator — Collaborative Neuroscience Network
Locations (1):
- Collaborative Neuroscience Network, Long Beach, California, United States